CLINICAL TRIAL: NCT06647420
Title: The Effect of Sedative and Stimulative Music Listening on State-Anxiety, Heart Rate, and Galvanic Skin Response in Nursing Students
Brief Title: The Effect of Music Listening on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Teresa Lesiuk, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20241018
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-10

CONDITIONS: Stress; Physiological Stress
Keywords: Heart rate; Skin conductance; Music

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sedative music followed by stimulative music group (Experimental): The participants in this group will receive sedative music followed by stimulative music for up to 25 minutes each. Session two will occur two days after session one.
  Interventions: Behavioral: Sedative Music; Behavioral: Stimulative Music
- Stimulative music followed by sedative music group (Experimental): The participants in this group will receive stimulative music followed by sedative music for up to 25 minutes each. Session two will occur two days after session one.
  Interventions: Behavioral: Sedative Music; Behavioral: Stimulative Music

INTERVENTIONS:
Behavioral: Sedative Music — The participants will come twice in person and listen to 9 minutes of sedative music.
Behavioral: Stimulative Music — The participants will come twice in person and listen to 9 minutes of stimulative music.

SUMMARY:
The purpose of this study is to explore the effect of sedative and stimulative music listening on physiological responses among nursing students.

ELIGIBILITY:
Inclusion criteria:

* a senior, junior, or second-semester sophomore in the traditional undergraduate Bachelor of Science in Nursing (BSN) program
* a student in the accelerated BSN program

Exclusion criteria:

•self-reported hearing impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate | baseline, up to 12 minutes
  Heart rate will be measured using the Polar Verity Sense Optical Heart Rate Sensor in beats per minute (bpm)
Change in Skin Conductance | baseline, up to 12 minutes
  Skin conductance will be measured using the NeuLog Galvanic Skin Response (GSR) in micro Siemens (µS).
Change in Anxiety Level | baseline, up to 12 minutes
  The Six Item State-Trait Anxiety Inventory includes six statements that are rated on a 4-point Likert scale (1=Not at all, 2=Somewhat, 3=Moderately so, 4=Very much). The scale will measure current feelings of anxiety.

SECONDARY OUTCOMES:
The Degree of Stress Experienced by A Nursing Student measured by the Perceived Stress Scale for Nursing Students (PSS) Likert Scale | up to 5 minutes
  The PSS consists of 29 items that are rated on a 5-point Likert scale (1=Never, 2=Seldom, 3=Sometimes, 4=Often, 5=Always). The PSS measures the degree of stress experienced by a nursing student based on stressful factors relevant to the demanding nursing curriculum.
Liking Song Scale (4-point Likert Scale) | up to 5 minutes
  Each music playlist will consist of three songs. The participant will rate how much the participant liked each of the three songs on a 4-point Likert scale (1=Not at all, 2=Somewhat, 3=Moderately so, 4=Very much).
Familiarity Song Scale (Rating scale) | up to 5 minutes
  Each music playlist will consist of three songs. The participant will indicate how familiar the participant is with each of the three songs on a rating scale (0=No, 1= I'm not sure, 2=Yes). The results of each song will be added to represent a quasi-continuous variable for how familiar the participant was with the music playlist as a whole.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Lesiuk, PhD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - University of Miami School of Nursing and Health Studies, Coral Gables, Florida
  - University of Miami, Coral Gables, Florida
  - Weeks Music Library and Technology Center, Coral Gables, Florida

IPD SHARING:
Plan to Share IPD: No